CLINICAL TRIAL: NCT01905930
Title: A Prospective, Randomized, Multi-Center, Post-Approval Clinical Trial Evaluating the Long-Term (7 Year) Safety and Effectiveness of the PCM® Cervical Disc
Brief Title: Post-Approval Clinical Trial of the PCM® Cervical Disc
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUVA-PCM-1101
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Radiculopathy; Myelopathy
MeSH Terms: conditions — Radiculopathy; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCM Cervical Disc (Experimental): Patients enrolled in the IDE clinical study and treated with the PCM Cervical Disc to treat degenerated cervical discs and neurological symptoms at one level from C3 to T1
  Interventions: Device: PCM Cervical Disc
- Ant. Cervical Discectomy & Fusion(ACDF) (Active Comparator): Patients enrolled in the IDE clinical study and treated with an anterior cervical discectomy and fusion (ACDF) using a cervical plate and bone graft in patients with degenerated cervical discs and neurological symptoms at one level from C3 to T1
  Interventions: Device: Anterior Cervical Discectomy and Fusion (ACDF)

INTERVENTIONS:
Device: PCM Cervical Disc — Patients enrolled in the IDE clinical study and treated with the PCM Cervical Disc to treat degenerated cervical discs and neurological symptoms at one level from C3 to T1
  Arms: PCM Cervical Disc
Device: Anterior Cervical Discectomy and Fusion (ACDF) — Patients enrolled in the IDE clinical study and treated with an anterior cervical discectomy and fusion (ACDF) using a cervical plate and bone graft in patients with degenerated cervical discs and neurological symptoms at one level from C3 to T1
  Arms: Ant. Cervical Discectomy & Fusion(ACDF)

SUMMARY:
On October 26, 2012, the FDA granted Premarket Approval (PMA) for the PCM Cervical Disc. PCM Cervical Disc is indicated for use in skeletally mature patients for reconstruction of a degenerated cervical disc at one level from C3-C4 to C6-C7 following single-level discectomy for intractable radiculopathy (arm pain and/or a neurological deficit), with or without neck pain, or myelopathy due to a single-level abnormality localized to the disc space, and manifested by at least one of the following conditions confirmed by radiographic imaging (CT, MRI, X-rays): herniated nucleus pulposus, spondylosis (defined by the presence of osteophytes), and/or visible loss of disc height as compared to adjacent levels.

The purpose of this post-approval study is to evaluate the long-term (7 year) safety and effectiveness of the PCM Cervical Disc.

DETAILED DESCRIPTION:
A prospective, multi-center, post approval study with concurrent control group consisting of those patients that were enrolled and did not fail in the PCM Cervical Disc IDE clinical study and will to give consent to participate.

All of the PCM IDE investigational sites who have active patients will be chosen to participate in this study. All patients who are actively participating in the pivotal IDE study will be asked to participate in this study.

The study consists of follow-up periods only. The follow-up period will last for seven years from each patient's surgery date.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the PCM Cervical Disc IDE clinical study
* Patients willing and able to give informed consent

Exclusion Criteria:

* Patients considered failure during the PCM Cervical Disc IDE clinical study
* Patients who were withdrawn during the PCM Cervical Disc IDE clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Individual Patient Overall Success | 7 years
  * Improvement of at least 20% on the Neck Disability Index (NDI) at 7 years compared to baseline
  * No device failures requiring revision, reoperation, removal or supplemental fixation
  * No major complications such as vascular or neurological injury
  * Radiographic success

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Spine Group Beverly Hills, Beverly Hills, California
  - Denver Spine, Greenwood Village, Colorado
  - Midwest Orthopedic Associates at Rush, Chicago, Illinois
  - Chicago Back Institute, Chicago, Illinois
  - Goodman Campbell Brain and Spine, Indianapolis, Indiana
  - Towson Orthopedic Associates, Towson, Maryland
  - Wm. Beaumont Hospital, Southfield, Michigan
  - Columbia Orthopedic Research, Columbia, Missouri
  - Buffalo Spine Surgery, Lockport, New York
  - Institute for Spine Care, Syracuse, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - Neuroscience Specialists, Oklahoma City, Oklahoma
  - The Rothman Institute, Philadelphia, Pennsylvania
  - Scott and White Memorial Hospital, Temple, Texas
  - Virginia Brain and Spine, Winchester, Virginia
  - Olympia Othopaedic Associates, Olympia, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - NeuroSpine Center of Wisconsin, Appleton, Wisconsin

REFERENCES:
- See also: Related Info — http://www.nuvasive.com